CLINICAL TRIAL: NCT01539746
Title: Use of the Self-Expanding Medtronic CoreValve Prosthesis Without Predilation in Patients With Severely IMPaired Left-VentrIcular Ejection Fraction for TAVI Trial - The SIMPLIFy TAVI Trial
Brief Title: Transcatheter Aortic Valve Implantation Without Predilation
Acronym: SIMPLIFy TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Georg Nickenig, Director, Department of Medicine II, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMPLIFy TAVI Trial
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Aortic Stenosis; Left Ventricular Function Systolic Dysfunction; High-risk Patients; Transcatheter Aortic Valve Implantation
Keywords: Aortic stenosis; Transcatheter aortic valve implantation; TAVI; Predilation; Balloon valvuloplasty; BAV; CoreValve
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAVI without predilation (Experimental)
  Interventions: Procedure: TAVI without BAV
- Standard TAVI procedure (Active Comparator)
  Interventions: Procedure: TAVI standard procedure

INTERVENTIONS:
Procedure: TAVI without BAV — Avoidance of balloon valvuloplasty (BAV) of the native aortic valve before valve deployment
  Arms: TAVI without predilation
Procedure: TAVI standard procedure — TAVI standard procedure including BAV before valve deployment
  Arms: Standard TAVI procedure

SUMMARY:
The purpose of this study is to demonstrate that the avoidance of balloon valvuloplasty for predilation of the native aortic valve is associated with a reduction of the composite primary endpoint in TAVI patients with severely impaired left-ventricular ejection fraction (LVEF ≤35%).

DETAILED DESCRIPTION:
Transcatheter aortic valve implantation (TAVI) has evolved as an alternative to surgical aortic valve replacement (SAVR) with now more than 50,000 implantations in patients with symptomatic severe aortic stenosis, who were considered to be at very high or prohibitive operative risk. Before deployment of transcatheter heart valves (THV), current medical practice requires right-ventricular rapid burst pacing (>180 bpm) with induction of a functional cardiac arrest for up to 30 seconds for balloon aortic valvuloplasty (BAV). This step is thought to be necessary to predilate the native aortic valve and to facilitate an accurate positioning of the THV. However, BAV has been shown to have numerous detrimental effects: i) the functional cardiac arrest induced by rapid pacing for BAV leads to transient coronary, cerebral, and renal ischemia. ii) In patients with impaired left ventricular ejection fraction, prolonged cardiac depression after rapid pacing is observed and may result in hemodynamic failure and systemic inflammatory response syndrome (SIRS), which are both associated with a high peri-procedural mortality. iii) BAV has been identified as a major source of embolization of thrombotic and valvular material and increases the risk for coronary obstruction with subsequent myocardial infarction and stroke. iv) the local trauma in the left-ventricular outflow tract caused by BAV contributes to conduction disturbances with the need for permanent pacemaker implantation after TAVI.

A non-randomized pilot study by Grube et al. (JACC Interventions 2011) has recently shown that TAVI without BAV is feasible and safe, since self-expanding THV are able to "dilate" the stenosed aortic valve through the radial forces of the self-expanding nitinol frame, in which the prosthesis is mounted. According to the mentioned study, omitting BAV allows the delivery of the THV in a controlled fashion without hemodynamic compromise of the patient.

Patients with LVEF≤35% will be randomized (like the flip of a coin) to TAVI without BAV (experimental group) or TAVI with BAV for predilation (control group).

ELIGIBILITY:
Inclusion Criteria:

* LVEF ≤35%
* Aortic valve stenosis with an aortic valve area <1 cm2 (<0,6 cm3/m2)
* Males or females at least 18 years of age
* Logistic EuroSCORE ≥15% and age ≥75 years or if age <75 years: logistic EuroSCORE ≥20% and/or a significant contraindication for open heart surgery (e.g., porcelain aorta or severe COPD)
* Signed informed consent

Exclusion Criteria:

* Patients with a device regulating the heart rhythm by pacing (e.g. pacemaker, resynchronization device, implanted defibrillator)
* Patients with a pre-existing class I or class II indication for new pacemaker implantation according to the 2007 ESC guidelines
* Lack of written informed consent, severe mental disorder, drug/alcohol addiction
* Life expectancy < 1 year
* Hypersensitivity or contraindication to acetyl salicyl acid, heparin, ticlopidine, clopidogrel, nitinol or sensitivity to contrast media that cannot be adequately premedicated
* Recent myocardial infarction (STEMI within the last 3 months)
* Left ventricular or atrial thrombus by echocardiography
* Uncontrolled atrial fibrillation
* Mitral or tricuspidal valvular insufficiency (> grade II)
* Previous aortic valve replacement with mechanical valve
* Evolutive or recent cerebrovascular event (within the last 3 months)
* Vascular conditions that make insertion and endovascular access to the aortic valve impossible
* Symptomatic carotid or vertebral arterial narrowing (>70%) disease
* Abdominal or thoracic aortic aneurysm in the path of the delivery system
* Bleeding diathesis or coagulopathy or patient refusing blood transfusion
* Active gastritis or peptic ulcer disease
* Severely impaired renal function, GFR < 30 ml/min
* Participation in another drug or device study that would jeopardize the appropriate analysis of end-points of this study.
* High probability of non-adherence to the follow-up requirements (due to social, psychological or medical reasons)
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-01-09 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Primary composite efficacy endpoint | 30 days after TAVI
  Occurrence of all-cause mortality, stroke, non-fatal myocardial infarction, acute kidney injury, or pacemaker implantation at 30 days after TAVI.

SECONDARY OUTCOMES:
Cardiovascular & all-cause mortality | 6 months, 12 months after TAVI
Major/minor stroke | 6 months, 12 months after TAVI
Myocardial infarction | 6 months, 12 months after TAVI
conduction disturbances and pacemaker implantation rate | 6 months, 12 months after TAVI
Acute kidney injury | 6 months, 12 months after TAVI
Rate of postdilation | 30 days, 6 months, 12 months after TAVI
Transvalvular mean gradient as assessed by echocardiography | 30 days, 6 months, 12 months after TAVI
Re-hospitalization for symptoms of cardiac/valve-related decompensation | 30 days, 6 months, 12 months after TAVI
Severity of periprosthetic aortic regurgitation (AR) as assessed by echocardiography, angiography, and hemodynamic measurements (AR index) | 30 days, 6 months, 12 months after TAVI
Life-threatening/major/minor bleeding | 30 days, 6 months, 12 months after TAVI
Vascular access complications | 30 days, 6 months, 12 months after TAVI
Repeat procedure for valve-related dysfunction (surgical or interventional therapy) | 30 days, 6 months, 12 months after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nickenig, MD, Principal Investigator — Department of Medicine II, University Hospital Bonn; Jan-Malte Sinning, MD, Study Director — Department of Medicine II, University Hospital Bonn
Locations (6):
- Germany (6):
  - Department of Medicine II - Cardiology, University Hospital Bonn, Bonn
  - Department of Cardiology, University Hospital Düsseldorf, Düsseldorf
  - West German Heart Center, University Hospital Essen, Essen
  - Department of Medicine III - Cardiology, University Hospital Heidelberg, Heidelberg
  - Department of Cardiology, Hospital Barmherzige Brüder Trier, Trier
  - Department of Medicine III - Cardiology, University Hospital Tübingen, Tübingen

REFERENCES:
- [Background] Grube E, Naber C, Abizaid A, Sousa E, Mendiz O, Lemos P, Kalil Filho R, Mangione J, Buellesfeld L. Feasibility of transcatheter aortic valve implantation without balloon pre-dilation: a pilot study. JACC Cardiovasc Interv. 2011 Jul;4(7):751-7. doi: 10.1016/j.jcin.2011.03.015. PMID 21777882
- [Background] Leon MB, Piazza N, Nikolsky E, Blackstone EH, Cutlip DE, Kappetein AP, Krucoff MW, Mack M, Mehran R, Miller C, Morel MA, Petersen J, Popma JJ, Takkenberg JJ, Vahanian A, van Es GA, Vranckx P, Webb JG, Windecker S, Serruys PW. Standardized endpoint definitions for Transcatheter Aortic Valve Implantation clinical trials: a consensus report from the Valve Academic Research Consortium. J Am Coll Cardiol. 2011 Jan 18;57(3):253-69. doi: 10.1016/j.jacc.2010.12.005. Epub 2011 Jan 7. PMID 21216553
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Sinning JM, Scheer AC, Adenauer V, Ghanem A, Hammerstingl C, Schueler R, Muller C, Vasa-Nicotera M, Grube E, Nickenig G, Werner N. Systemic inflammatory response syndrome predicts increased mortality in patients after transcatheter aortic valve implantation. Eur Heart J. 2012 Jun;33(12):1459-68. doi: 10.1093/eurheartj/ehs002. Epub 2012 Jan 26. PMID 22285582
- [Background] Nuis RJ, Van Mieghem NM, Schultz CJ, Tzikas A, Van der Boon RM, Maugenest AM, Cheng J, Piazza N, van Domburg RT, Serruys PW, de Jaegere PP. Timing and potential mechanisms of new conduction abnormalities during the implantation of the Medtronic CoreValve System in patients with aortic stenosis. Eur Heart J. 2011 Aug;32(16):2067-74. doi: 10.1093/eurheartj/ehr110. Epub 2011 May 28. PMID 21622979
- [Background] Kahlert P, Erbel R. Transcatheter aortic valve implantation in the era after commercialization: quo vadis in the real world? Circulation. 2011 Jan 25;123(3):239-41. doi: 10.1161/CIRCULATIONAHA.110.004713. Epub 2011 Jan 10. No abstract available. PMID 21220739
- [Background] Ghanem A, Muller A, Nahle CP, Kocurek J, Werner N, Hammerstingl C, Schild HH, Schwab JO, Mellert F, Fimmers R, Nickenig G, Thomas D. Risk and fate of cerebral embolism after transfemoral aortic valve implantation: a prospective pilot study with diffusion-weighted magnetic resonance imaging. J Am Coll Cardiol. 2010 Apr 6;55(14):1427-32. doi: 10.1016/j.jacc.2009.12.026. Epub 2010 Feb 24. PMID 20188503
- [Background] Drews T, Pasic M, Buz S, Unbehaun A, Dreysse S, Kukucka M, Mladenow A, Hetzer R. Transcranial Doppler sound detection of cerebral microembolism during transapical aortic valve implantation. Thorac Cardiovasc Surg. 2011 Jun;59(4):237-42. doi: 10.1055/s-0030-1250495. Epub 2011 Mar 25. PMID 21442580
- [Background] Sinning JM, Ghanem A, Steinhauser H, Adenauer V, Hammerstingl C, Nickenig G, Werner N. Renal function as predictor of mortality in patients after percutaneous transcatheter aortic valve implantation. JACC Cardiovasc Interv. 2010 Nov;3(11):1141-9. doi: 10.1016/j.jcin.2010.09.009. PMID 21087750